CLINICAL TRIAL: NCT00308828
Title: Prevalence of Osteoporosis in Hemodialysis Patients and Relevance With Renal Bone Disease
Brief Title: The Prevalence of Osteoporosis in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Papageorgiou General Hospital (Other)
Responsible Party: Efstathios Mitsopoulos, Papageorgiou General Hospital, Thessaloniki, Greece
Other Study IDs: 47/31-1-2005
Record Dates: First submitted 2006-03-29; First posted 2006-03-30 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
The purpose of this study is to determine the prevalence and severity of osteoporosis in hemodialysis patients and to evaluate potential correlations with renal bone disease indices

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis
* Age > 18-year old

Exclusion Criteria:

* Prior specific osteoporosis treatment except vitamin D and calcium supplement administration; active malignancy
* Recent pregnancy
* Immobilization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Mitsopoulos, MD, Principal Investigator — Papageorgiou General Hospital
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Greece